CLINICAL TRIAL: NCT03724513
Title: High Altitude Area- A Risk Factor For Gastric Perforation?
Status: Completed | Type: Observational
Sponsor: ADITYA PAWAR (Other Government)
Responsible Party: Sponsor-Investigator, ADITYA PAWAR, Principal Investigator, 403 Military Field Hospital, India
Organization: 403 Military Field Hospital, India (Other Government)
Other Study IDs: 403HAAPPU
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Gastric Perforation
Keywords: High Altitude; Gastric Antrum Perforation; Mucosal Atrophy; Intra Luminal Pressure
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an original case series on soldiers evacuated from HAA(High Altitude Area) over last one year(Sept 2017- Aug 2018) , of which 100% cases were found to have gastric antrum perforation. This is a deviation from the usual trend that is being noted in Indian subcontinent where duodenal perforations are commonest.

DETAILED DESCRIPTION:
INTRODUCTION : This is an original case series on soldiers evacuated from HAA(High Altitude Area) over last one year(Sept 2017- Aug 2018) , of which 100% cases were found to have gastric antrum perforation. This is a deviation from the usual trend that is being noted in Indian subcontinent where duodenal perforations are commonest.

DISCUSSION : High altitude associated dyspepsia is a common phenomenon and some studies done in high altitude population have recorded high incidence of antral gastritis and mucosal atrophy on histo-pathological evaluation. This is also supported by high incidence of H.pylori infection. The presence of atrophic gastric mucosa associated with antral gastritis, when exposed to hypobaric hypoxemic conditions faced by soldiers posted to heights above 15000ft , may leads to increased intra-luminal pressure and ischemia which probably predisposes individuals for gastric antrum perforations.

CONCLUSION : This is a relatively untouched topic as we have not found studies on high altitude related gastric perforations and probably this is the first case series of its kind. The acknowledgement of this phenomenon may pave way for further studies for defining the role of high altitude in gastric perforations.

ELIGIBILITY:
Inclusion Criteria:

* Individuals located in High Altitude Area (>10,000ft).
* presented as perforation peritonitis.
* intra-operatively found to be perforated peptic ulcers.

Exclusion Criteria:

* Not located in High Altitude Area.
* intra-operatively perfoarations sites other then stomach and duodenum.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Young soldiers located in High Altitude Area
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Assessment of site of perforated peptic ulcers by intra-operative observation in cases evacuated from High Altitude Area. | 1 year
  Study aims at recording the site of perforated peptic ulcers in cases being evacuated in individuals posted at High Altitude Area.

CONTACTS AND LOCATIONS:
Overall Officials: Aditya Pawar, MS, Principal Investigator — 403 MILITARY FIELD HOSPITAL
Locations (1):
- 403 Military Field Hospital, Leh, Jammu and Kashmir, India

IPD SHARING:
Plan to Share IPD: No